CLINICAL TRIAL: NCT00965874
Title: Low Versus High Dose Magnesium Sulfate in the Early Management of Rapid Atrial Fibrillation : Randomised Controlled Double Blind Study (LOMAGHI Study)
Brief Title: Low Versus High Dose Magnesium Sulfate in the Early Management of Rapid Atrial Fibrillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LOMAGHI
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Atrial Fibrillation
Keywords: Rapid Atrial Fibrillation; Magnesium Sulfate; Cardiac arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Magnesium Sulfate high dose infusion (Experimental): 9 g Magnesium sulfate infusion over 30 minutes
  Interventions: Drug: Magnesium Sulfate high dose
- Magnesium Sulfate low dose infusion (Active Comparator): 4.5 magnesium sulfate infusion over 30 minutes
  Interventions: Drug: Magnesium Sulfate low dose
- placebo (Placebo Comparator): serum salin
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Magnesium Sulfate high dose — 9 g infusion once during 30 minutes
  Other Names: Magnesium Sulfate
  Arms: Magnesium Sulfate high dose infusion
Drug: Magnesium Sulfate low dose — 4.5 g magnesium sulfate infusion
  Other Names: Magnesium Sulfate
  Arms: Magnesium Sulfate low dose infusion
Drug: Placebos — serum salin
  Arms: placebo

SUMMARY:
Objective:

To assess the efficacy and the safety of high (9g) and low dose (4.5g) of MgS in the immediate treatment of rapid AF.

DETAILED DESCRIPTION:
Introduction:

Atrial fibrillation (AF) is a potentially life-threatening cardiac arrhythmia and a frequent chief complaint in emergency departments (ED). It is an important concern for a substantial proportion of people worldwide. According to the Rotterdam study, the prevalence of AF among individuals aged between 55 to 59 years is estimated at 1.1 for 1000 persons/year and 20.7 for individuals between 80 and 84 years. Given current adult advanced cardiac life support (ACLS), the immediate clinical objective in rapid AF is to achieve ventricular rate control. Digoxin, beta blockers and calcium channel antagonists are the most widely used agents for the emergent treatment of rapid AF. However, their effect is limited because only half of the patients will acutely respond to the first intention treatment. Several studies showed that the magnesium sulfate (MgS) is beneficial in the control of the rate and the rhythm of AF. In addition, hypomagnesemia is present among patients having AF in 20 to 53% of the cases . The association of hypomagnesemia and AF is common after a cardiac surgery and the prophylactic administration of MgS could be useful in post-operative AF .

The last meta analysis published in 2007 showed that the MgS is as well efficient in rate control (OR = 1.96) as in rhythm control (OR = 1.60) of AF. However most studies included in this meta analysis were conducted on limited number of patients (303 patients included for rate control outcome analysis and 376 for rhythm control). Consequently we need further randomized controlled studies to establish definitively the efficacy and the safety of MgS in the early management of rapid AF.

Objective:

To assess the efficacy and the safety of high (9g) and low dose (4.5g) of MgS in the immediate treatment of rapid AF.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to ED with rapid AF (Heart rate >120 bpm).

Exclusion Criteria:

* Unstable hemodynamic state.
* Renal insufficiency (creatinemia> 180 µmol/l).
* Allergy to MgS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
HR <90 bpm or 20% reduction from baseline at 24 hours | 24 hours

SECONDARY OUTCOMES:
Arterial hypotension Bradycardia (HR <45 bpm) Other (chest pain, allergic reaction……) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: nouira semir, MD, Principal Investigator — University of Monastir
Locations (1):
- University Hospital of Monastir, Monastir, Monstir, Tunisia

IPD SHARING:
Plan to Share IPD: Yes